CLINICAL TRIAL: NCT02940886
Title: A Phase III, Randomised, Open-label, Comparative Safety and Efficacy Trial of Intravenous Iron Isomaltoside/Ferric Derisomaltose (Monofer®/Monoferric®) and Iron Sucrose in Subjects With Iron Deficiency Anemia (FERWON-IDA)
Brief Title: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose for the Treatment of Iron Deficiency Anemia (IDA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-IDA-03
Record Dates: First submitted 2016-09-27; First posted 2016-10-21 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-01

CONDITIONS: Iron Deficiency Anaemia; Iron Deficiency Anemia
Keywords: Iron Deficiency Anaemia; Iron Deficiency Anemia; IDA; Intravenous iron replacement therapy; Iron isomaltoside; Ferric derisomaltose; Monofer; Monoferric; Monover; Monofar; Monoferro
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — iron isomaltoside 1000; ferric derisomaltose; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iron isomaltoside/ferric derisomaltose (Experimental): Administered IV
  Interventions: Drug: Iron isomaltoside/ferric derisomaltose
- Iron sucrose (Active Comparator): Administered IV
  Interventions: Drug: Iron sucrose

INTERVENTIONS:
Drug: Iron isomaltoside/ferric derisomaltose — Iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) was the test product in this trial.
  The dose of iron isomaltoside/ferric derisomaltose for the individual subject was set to 1000 mg. The dose was diluted in 100 mL 0.9 % sodium chloride (100 mL bags) and administered as a single IV infusion over approximately 20 minutes.
  Other Names: Monofer®, Monoferric®, Monover®, Monofar®, Monoferro®
  Arms: Iron isomaltoside/ferric derisomaltose
Drug: Iron sucrose — Iron sucrose (Venofer®; 20 mg elemental iron/mL) was the comparator in this trial.
  Iron sucrose was administered as 200 mg undiluted IV injections over approximately 2-5 minutes and repeated according to standard practice or physician choice up to a maximum of five times within the first two weeks starting at baseline. A cumulative dose of 1000 mg was recommended.
  Other Names: Venofer®
  Arms: Iron sucrose

SUMMARY:
Evaluate safety and efficacy of iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®) compared with iron sucrose (Venofer®), in subjects diagnosed with IDA.

DETAILED DESCRIPTION:
IDA is highly prevalent condition in subjects with cancer and gastrointestinal diseases such as inflammatory bowel diseases, menstruating or pregnant women, and subjects who have undergone bariatric procedure or surgery. IDA can have a substantial medical and quality of life (QoL) burden. Treatment of subjects diagnosed with IDA includes controlling the bleeding and replenishing lost iron.

This study was designed to evaluate the safety and efficacy of iron isomaltoside/ferric derisomaltose compared with iron sucrose in subjects diagnosed with IDA. In a subfraction of 35 subjects treated with iron isomaltoside/ferric derisomaltose, ECG and iron will be frequently measured.

The study subjects received either a single intravenous (IV) dose of iron isomaltoside/ferric derisomaltose (1000 mg at baseline) or iron sucrose (200 mg IV injections at baseline and repeated according to standard practice or physician choice up to a maximum of five times within the first two weeks starting at baseline; a cumulative dose of 1000 mg was recommended). The study subjects were monitored for up to 8 weeks from baseline.

ELIGIBILITY:
Inclusion criteria includes:

1. Men or women ≥ 18 years
2. Subjects having IDA caused by different etiologies
3. Subjects with intolerance to oral iron therapy or a need for rapid repletion of iron stores:
4. Haemoglobin (Hb) ≤ 11 g/dL
5. Transferrin Saturation (TSAT) < 20 %
6. S-ferritin < 100 ng/mL
7. Willingness to participate and signing the informed consent form

Exclusion Criteria includes :

1. Anemia predominantly caused by factors other than IDA
2. Hemochromatosis or other iron storage disorders
3. Previous serious hypersensitivity reactions to any IV iron compound
4. Erythropoiesis stimulating agent (ESA) treatment
5. Prior to screening or during the trial period; has or will be treated with a red blood cell transfusion, radiotherapy, and/or chemotherapy
6. Will require a surgical procedure that necessitated general anesthesia prior to screening or during the trial period
7. Alanine aminotransferase and/or aspartate aminotransferase > 3 times upper limit of normal
8. Required dialysis for treatment of chronic kidney disease (CKD)
9. Alcohol or drug abuse within the past 6 months
10. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1512 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacosmos A/S Clinical and Non-clinical Research, Study Director — Pharmacosmos A/S
Locations (96):
- United States (96):
  - Pharmacosmos Investigational Site, Birmingham, Alabama
  - Pharmacosmos Investigational Site, Dothan, Alabama
  - Pharmacosmos Investigational Site, Guntersville, Alabama
  - Pharmacosmos Investigational Site, Phoenix, Arizona
  - Pharmacosmos Investigational Site, Little Rock, Arkansas
  - Pharmacosmos Investigational Site, Foothill Ranch, California
  - Pharmacosmos Investigational Site 1, La Mesa, California
  - Pharmacosmos Investigational Site 2, La Mesa, California
  - Pharmacosmos Investigational Site, Long Beach, California
  - Pharmacosmos Investigational Site, National City, California
  - Pharmacosmos Investigational Site 1, Northridge, California
  - Pharmacosmos Investigational Site 2, Northridge, California
  - Pharmacosmos Investigational Site, Oceanside, California
  - Pharmacosmos Investigational Site, Quartz Hill, California
  - Pharmacosmos Investigational Site, Rialto, California
  - Pharmacosmos Investigational Site, Riverside, California
  - Pharmacosmos Investigational Site, San Diego, California
  - Pharmacosmos Investigational Site, San Marcos, California
  - Pharmacosmos Investigational Site, Whittier, California
  - Pharmacosmos Investigational Site, Plainville, Connecticut
  - Pharmacosmos Investigational Site, Aventura, Florida
  - Pharmacosmos Investigational Site, Boynton Beach, Florida
  - Pharmacosmos Investigational Site 1, Doral, Florida
  - Pharmacosmos Investigational Site 2, Doral, Florida
  - Pharmacosmos Investigational Site, Doral, Florida
  - Pharmacosmos Investigational Site, Fort Lauderdale, Florida
  - Pharmacosmos Investigational Site, Hialeah, Florida
  - Pharmacosmos Investigational Site, Hollywood, Florida
  - Pharmacosmos Investigational Site, Jacksonville, Florida
  - Pharmacosmos Investigational Site, Kissimmee, Florida
  - Pharmacosmos Investigational Site, Lake City, Florida
  - Pharmacosmos Investigational Site, Lake Worth, Florida
  - Pharmacosmos Investigational Site, Miami, Florida
  - Pharmacosmos Investigational Site 1, Miami, Florida
  - Pharmacosmos Investigational Site 2, Miami, Florida
  - Pharmacosmos Investigational Site 1, Miami Lakes, Florida
  - Pharmacosmos Investigational Site 2, Miami Lakes, Florida
  - Pharmacosmos Investigational Site, Miami Lakes, Florida
  - Pharmacosmos Investigational Site 1, Naples, Florida
  - Pharmacosmos Investigational Site 2, Naples, Florida
  - Pharmacosmos Investigational Site, Palmetto Bay, Florida
  - Pharmacosmos Investigational Site, Plantation, Florida
  - Pharmacosmos Investigational Site, West Palm Beach, Florida
  - Pharmacosmos Investigational Site, Champaign, Illinois
  - Pharmacosmos Investigational Site, Joliet, Illinois
  - Pharmacosmos Investigational Site, Palos Heights, Illinois
  - Pharmacosmos Investigational Site, Terre Haute, Indiana
  - Pharmacosmos Investigational Site, Wichita, Kansas
  - Pharmacosmos Investigational Site, Owensboro, Kentucky
  - Pharmacosmos Investigational Site, Baton Rouge, Louisiana
  - Pharmacosmos Investigational Site, Marrero, Louisiana
  - Pharmacosmos Investigational Site, Metairie, Louisiana
  - Pharmacosmos Investigational Site, New Orleans, Louisiana
  - Pharmacosmos Investigational Site, Shreveport, Louisiana
  - Pharmacosmos Investigational Site, Bethesda, Maryland
  - Pharmacosmos Investigational Site, Hagerstown, Maryland
  - Pharmacosmos Investigational Site, Towson, Maryland
  - Pharmacosmos Investigational Site, Fall River, Massachusetts
  - Pharmacosmos Investigational Site, Grand Rapids, Michigan
  - Pharmacosmos Investigational Site, Saginaw, Michigan
  - Pharmacosmos Investigational Site, Troy, Michigan
  - Pharmacosmos Investigational Site, Florissant, Missouri
  - Pharmacosmos Investigational Site, Omaha, Nebraska
  - Pharmacosmos Investigational Site, Las Vegas, Nevada
  - Pharmacosmos Investigational Site, Neptune City, New Jersey
  - Pharmacosmos Investigational Site, Plainsboro, New Jersey
  - Brooklyn, New York
  - Pharmacosmos Investigational Site 1, East Setauket, New York
  - Pharmacosmos Investigational Site 2, East Setauket, New York
  - Pharmacosmos Investigational Site, New York, New York
  - Pharmacosmos Investigational Site, Wilmington, North Carolina
  - Pharmacosmos Investigational Site, Beavercreek, Ohio
  - Pharmacosmos Investigational Site, Canton, Ohio
  - Pharmacosmos Investigational Site, Centerville, Ohio
  - Pharmacosmos Investigational Site, Cincinnati, Ohio
  - Pharmacosmos Investigational Site, Columbus, Ohio
  - Pharmacosmos Investigational Site, Norman, Oklahoma
  - Pharmacosmos Investigational Site, Tulsa, Oklahoma
  - Pharmacosmos Investigational Site, Jenkintown, Pennsylvania
  - Pharmacosmos Investigational Site, Columbia, South Carolina
  - Pharmacosmos Investigational Site, Myrtle Beach, South Carolina
  - Pharmacosmos Investigational Site, Chattanooga, Tennessee
  - Pharmacosmos Investigational Site, Franklin, Tennessee
  - Pharmacosmos Investigational Site, Knoxville, Tennessee
  - Pharmacosmos Investigational Site, Memphis, Tennessee
  - Pharmacosmos Investigational Site, Austin, Texas
  - Pharmacosmos Investigational Site, Baytown, Texas
  - Pharmacosmos Investigational Site, Beaumont, Texas
  - Pharmacosmos Investigational Site, Corsicana, Texas
  - Pharmacosmos Investigational Site, DeSoto, Texas
  - Pharmacosmos Investigational Site, Houston, Texas
  - Pharmacosmos Investigational Site, McAllen, Texas
  - Pharmacosmos Investigational Site, San Antonio, Texas
  - Pharmacosmos Investigational Site, Ogden, Utah
  - Pharmacosmos Investigational Site, Chesapeake, Virginia
  - Pharmacosmos Investigational Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Auerbach M, Henry D, Derman RJ, Achebe MM, Thomsen LL, Glaspy J. A prospective, multi-center, randomized comparison of iron isomaltoside 1000 versus iron sucrose in patients with iron deficiency anemia; the FERWON-IDA trial. Am J Hematol. 2019 Sep;94(9):1007-1014. doi: 10.1002/ajh.25564. Epub 2019 Jul 13. PMID 31243803
- [Result] Auerbach M and Lykke LL. A single infusion of iron isomaltoside 1000 allows a more rapid hemoglobin increment than multiple doses of iron sucrose with a similar safety profile in patients with iron deficiency anemia. Blood 2018 132:2334; doi: https://doi.org/10.1182/blood-2018-99-110199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 3108 subjects were screened and 1512 subjects were randomised in the trial.
Pre-assignment Details: Subjects who did not have a documented history of intolerance of oral iron for at least 1 month within the last 9 months had a run-in period. During the run-in period, the subject received oral iron for up to 1 month in order to document intolerance or lack of response to oral iron.Subjects were monitored for AEs indicative of iron intolerance.
Groups:
- Iron Isomaltoside/Ferric Derisomaltose: Iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) was the test product in this trial.
  Subjects received iron isomaltoside/ferric derisomaltose (Monofer®/Monoferric®; 100 mg/mL) as a single IV infusion of 1000 mg at the baseline visit.
- Iron Sucrose: Iron sucrose (Venofer®) was the comparator in this trial.
  Subjects received iron sucrose (Venofer®), 200 mg IV injection up to a maximum of 5 intravenous injections within the first 2 weeks, starting at baseline (a cumulative dose of 1000 mg was recommended).
Period: Overall Study
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Started | 1009 (Intention-to-treat analysis set included 1009 subjects, safety analysis set included 989 subjects.) | 503 (Intention-to-treat analysis set included 503 subjects, safety analysis set included 494 subjects.)
Safety Analysis Set | 989 | 494
Completed | 907 | 449
Not Completed | 102 | 54
Not completed — Adverse Event | 7 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 28 | 20
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 49 | 21
Not completed — Physician Decision | 9 | 4
Not completed — Sponsor decision | 0 | 1
Not completed — No treatment | 7 | 2
Not completed — Enrolment error | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Iron Isomaltoside/Ferric Derisomaltose: Iron isomaltoside/ferric derisomaltose, administered IV
- Iron Sucrose: Iron sucrose, administered IV
- Total: Total of all reporting groups
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose | Total
Number analyzed (Participants) | 1009 | 503 | 1512
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 902 | 440 | 1342
  >=65 years | 107 | 63 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (14.8) | 43.8 (14.4) | 44.0 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 892 | 456 | 1348
  Male | 117 | 47 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 387 | 205 | 592
  Not Hispanic or Latino | 622 | 298 | 920
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 8 | 4 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 484 | 223 | 707
  White | 504 | 264 | 768
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 5 | 9 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Arabic | 0 | 2 | 2
  Hispanic | 3 | 3 | 6
  Mix race (Black & White) | 3 | 0 | 3
  Caucasian | 0 | 1 | 1
  Haitian | 0 | 1 | 1
  Latino | 1 | 0 | 1
  Other (not declared) | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 1009 | 503 | 1512
Current smoker [Count of Participants; unit: Participants]
  YES | 133 | 80 | 213
  NO | 876 | 423 | 1299

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hb) From Baseline to Week 8
Description: Efficacy
  Evaluate the effect on the hemoglobin (Hb) level following treatment with iron isomaltoside/ferric derisomaltose vs iron sucrose in subjects with iron deficiency anaemia (IDA) .
  Response was defined as change from baseline in hemoglobin (Hb) to week 8, i.e. ability to increase Hb in subjects with IDA, when oral iron preparations were ineffective or could not be used or in whom the screening Hb measurement in Investigators' opinion were sufficiently low to require rapid repletion of iron stores.
Time Frame: Baseline to week 8
Population: Intention to treat (ITT). All randomised subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
g/dL | 2.49 [2.41 to 2.56] | 2.49 [2.38 to 2.59]
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Power: With N=1000 subjects in the iron isomaltoside/ferric derisomaltose treatment group and with N=500 subjects in the iron sucrose treatment group, assuming no difference between the treatment groups and assuming a common standard deviation (SD) of 1.5 g/dL, the power was 100% for demonstrating non-inferiority of the change in Hb from baseline to week 8, using a non-inferiority margin of -0.5 g/dL. The significance level was set to 5%; Test type: Non-Inferiority — Non-inferiority could be claimed if the lower bound of the 95% confidence interval (CI) was above -0.5 g/dL; Mean Difference (Final Values) = 0.00, 95% CI 2-sided [-0.13 to 0.13] — Mixed Model for Repeated Measurement was used for testing and included the fixed categorical effects of treatment, week, treatment-by-week interaction, strata, and the continuous covariates of baseline Hb and baseline Hb-by-week interaction

2. Primary Outcome: Incidence of Protocol-defined Serious or Severe Hypersensitivity Reactions
Description: Safety
  For this endpoint, the number of participants with serious or severe hypersensitivity reactions were evaluated. The hypersensitivity reactions that were included in the analysis were those that started on or after the first dose of randomised treatment (i.e. treatment emergent). The terms used to define hypersensitivity were those specified by the Standardised MedDRA Queries (SMQ) for hypersensitivity, plus four additional terms: loss of consciousness, seizure, syncope, unresponsiveness.
  The potential hypersensitivity AEs were adjudicated in a blinded fashion by an independent Clinical Endpoint Adjudication Committee (CEAC).
  Results show only those participants that had adjudicated and confirmed serious or severe hypersensitivity reactions.
Time Frame: Baseline to week 8
Population: Safety analysis set. All randomised subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 989 | 494
Participants | 3 | 2
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose; Power: With N=1000 subjects in the iron isomaltoside/ferric derisomaltose, the power was 88% to demonstrate that the upper bound of the 95% CI of the incidence of treatment-emergent serious and/or severe non-serious hypersensitivity AEs was less than 3%. The significance level was set to 5%; Test type: Other; 95% two-sided CI (iron isomaltoside) = 0.3, 95% CI 2-sided [0.06 to 0.88]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Risk difference between iron isomaltoside/ferric derisomaltose and iron sucrose was assessed for the individual trial with 95% Newcombe CI adjusted for stratum using the Cochran-Mantel-Haenszel method; Test type: Other; Risk Difference (RD) = -0.10, 95% CI 2-sided [-0.91 to 0.71]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Risk difference between iron isomaltoside/ferric derisomaltose and iron sucrose was assessed for the pooled FERWON-IDA and FERWON-NEPHRO trials (2008 subjects treated with iron isomaltoside/ferric derisomaltose and 1000 subjects treated with iron sucrose) with 95% Newcombe CI adjusted for stratum using the Cochran-Mantel-Haenszel method; Test type: Non-Inferiority — Non-inferiority can be claimed if the upper bound of the 95% CI is below 1.5 % point; Risk Difference (RD) = 0.10, 95% CI 2-sided [-0.57 to 0.48]

3. Secondary Outcome: Composite Cardiovascular Adverse Events (AEs)
Description: Safety
  Results show the composite cardiovascular adverse events (AEs), that started on or after the first dose of randomised treatment (i.e. treatment emergent) up to week 8.
  The reported potential cardiovascular AEs were adjudicated in a blinded fashion by an independent Clinical Endpoint Adjudication Committee (CEAC).
  The potential cardiovascular AEs included the following:
  * Death due to any cause
  * Non-fatal myocardial infarction
  * Non-fatal stroke
  * Unstable angina requiring hospitalisation
  * Congestive heart failure requiring hospitalisation or medical intervention
  * Arrhythmias
  * Hypertension
  * Hypotension
  Results show only those participants that had adjudicated and confirmed treatment-emergent composite cardiovascular AEs.
Time Frame: Baseline, week 1, 2, and 8
Population: Safety analysis set. All randomised subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 989 | 494
Participants | 8 | 6
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Adjudicated and confirmed treatment-emergent composite cardiovascular AEs. Any treatment emergent composite cardiovascular AEs were included in the statistical evaluation. The overall incidence of adjudicated and confirmed composite cardiovascular AEs was tabulated and compared between the treatment groups by a Fisher's exact test; Test type: Superiority; p = 0.5695, Fisher Exact

4. Secondary Outcome: Time to First Composite Cardiovascular Safety AE
Description: Safety
  Time to first composite cardiovascular AE was defined as the actual time in days from first dose of treatment until the date of the composite cardiovascular AE. For subjects not reporting a composite cardiovascular AE, the time was censored at the date of the last attended visit. Only the adjudicated and confirmed composite cardiovascular safety AEs, as judged by the CEAC, were considered for this endpoint.
  Time to first composite cardiovascular AE was defined as the actual time in days from first dose of treatment until the date of the composite cardiovascular AE. For subjects not reporting a composite cardiovascular AE, the time was censored at the date of the last attended visit.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: Safety analysis set. All randomised subjects who received at least one dose of the investigational product.
Measure: Median (95% Confidence Interval); unit: Week
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 989 | 494
Week | NA [NA to NA] — The number of adjudicated and confirmed composite cardiovascular safety AEs was too low (N=8) for estimation of median and 95 % CI. | NA [NA to NA] — The number of adjudicated and confirmed composite cardiovascular safety AEs was too low (N=6) for estimation of median and 95 % CI.
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; The time to first adjudicated and confirmed composite cardiovascular AEs was estimated using the Kaplan-Meier method and the hypothesis of no treatment difference was assessed by a log-rank test; Test type: Superiority; p = 0.3913, Log Rank

5. Secondary Outcome: S-phosphate <2 mg/dL at Any Time From Baseline to Week 1, 2, 4, and 8
Description: Safety
  Results show the number of subjects who had s-phosphate <2 mg/dL at any time from baseline to week 1, 2, 4, or 8.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: Safety analysis set. All randomised subjects who received at least one dose of the investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 989 | 494
Participants | 38 | 11

6. Secondary Outcome: Hb Concentration Increase of ≥2 g/dL From Baseline to Week 1, 2, 4, and 8
Description: Efficacy
  Results show responders to the treatment. A subject was considered a Hb responder to a certain week if an increase in Hb of at least 2 g/dL from baseline to the week in question was observed (week 1, 2, 4, and 8).
Time Frame: Baseline, week 1, 2, 4, and 8
Population: ITT. All randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
Participants
  Responder YES week 1: number analyzed (Participants) | 960 | 477
  Responder YES week 1 | 51 | 12
  Responder YES week 2: number analyzed (Participants) | 912 | 452
  Responder YES week 2 | 297 | 94
  Responder YES week 4: number analyzed (Participants) | 903 | 450
  Responder YES week 4 | 514 | 250
  Responder YES week 8: number analyzed (Participants) | 903 | 454
  Responder YES week 8 | 606 | 309
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Hb increase of ≥2 g/dL from baseline to week 1. Proportion of Hb responders to each week was analysed using a repeated measures logistic regression model with treatment, visit, strata, and treatment by visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.0077, Repeated measures logistic regressioin; Odds Ratio (OR) = 2.44, 95% CI 2-sided [1.27 to 4.72]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Hb increase of ≥2 g/dL from baseline to week 2. Proportion of Hb responders to each week was analysed using a repeated measures logistic regression model with treatment, visit, strata, and treatment by visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p < 0.0001, Repeated measures logistic regressioin; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.80 to 3.26]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 4 Hb increase of ≥2 g/dL from baseline to week 4. Proportion of Hb responders to each week was analysed using a repeated measures logistic regression model with treatment, visit, strata, and treatment by visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.1049, Repeated measures logistic regressioin; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.96 to 1.58]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 8 Hb increase of ≥2 g/dL from baseline to week 8. Proportion of Hb responders to each week was analysed using a repeated measures logistic regression model with treatment, visit, strata, and treatment by visit interaction as fixed effects and baseline value as covariate; Test type: Superiority; p = 0.7032, Repeated measures logistic regressioin; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.80 to 1.38]

7. Secondary Outcome: Time to Change in Hb Concentration ≥2 g/dL
Description: Efficacy
  Time to change in Hb concentration ≥2 g/dL. Subjects who achieved Hb concentration increase of ≥2 g/dL (from baseline to week 1, 2, 4, or 8).
  For responders, time to Hb response was defined as the scheduled time from baseline until the visit where the first Hb response was measured.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: ITT. All randomised subjects.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
Days | 28 [NA to NA] — The 95% Confidence Interval values for this treatment group could not be calculated due to insufficient number of events. | 28 [28 to 56]
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Time to Hb response was estimated using the Kaplan-Meier method and the hypothesis of no treatment difference was assessed by a 2-sided log-rank test; Test type: Superiority; p = 0.0880, Log Rank

8. Secondary Outcome: Hb Concentration of >12 g/dL at Any Time From Week 1 to Week 8
Description: Efficacy
  Hb concentration of >12 g/dL at any time from week 1 to week 8.
  Results show the number of participants who achieved Hb concentration of >12 g/dL at any time from week 1 to week 8.
Time Frame: Week 1 to week 8
Population: ITT. All randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 502
Participants | 484 | 225
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; The proportion of subjects who achieved a Hb level of >12 g/dL at any time from week 1 to week 8 was analysed using a logistic regression model with treatment and strata as fixed effects. The estimated treatment ratio of iron isomaltoside/ferric derisomaltose versus iron sucrose is presented with 95% CI and corresponding p-value; Test type: Superiority; p = 0.2420, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.92 to 1.41]

9. Secondary Outcome: Hb Concentration Increase of ≥2 g/dL at Any Time From Week 1 to Week 8
Description: Efficacy
  Results show the number of participants who achieved Hb concentration increase of ≥2 g/dL at any time from week 1 to week 8.
Time Frame: Week 1 to week 8
Population: ITT. All randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 502
Participants | 687 | 340
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; The proportion of subjects who achieved an increase in Hb concentration ≥2 g/dL at any time from week 1 to week 8 was analysed using a logistic regression model with treatment and strata as fixed effects. The estimated treatment ratio of iron isomaltoside/ferric derisomaltose versus iron sucrose was presented with 95% CI and corresponding p-value; Test type: Superiority; p = 0.8746, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.81 to 1.28]

10. Secondary Outcome: S-Ferritin Concentration of ≥100 ng/mL and Transferrin Saturation (TSAT) of 20-50% at Any Time From Week 1 to Week 8
Description: Efficacy
  Proportion of subjects reaching the composite endpoint of s-ferritin concentration ≥100 ng/mL and TSAT of 20-50% at any time from week 1 to 8.
Time Frame: Week 1 to week 8
Population: ITT. All randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 973 | 483
Participants | 680 | 164
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Proportion of subject who achieved a s-ferritin level of ≥100 ng/mL AND a TSAT of 20-50% at any time from week 1 to week 8 was analysed using a logistic regression model with treatment and strata as fixed effects. The estimated treatment ratio of iron isomaltoside/ferric derisomaltose versus iron sucrose is presented with 95% CI and corresponding p-value; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.52, 95% CI 2-sided [3.58 to 5.71]

11. Secondary Outcome: Change in Hb Concentration From Baseline to Week 1, 2, and 4
Description: Efficacy
  Change in Hb concentration from baseline to week 1, 2, and 4.
Time Frame: Baseline, week 1, 2, and 4
Population: ITT. All randomised subjects.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
g/dL
  Week 1: number analyzed (Participants) | 960 | 477
  Week 1 | 0.70 (0.85) | 0.47 (0.69)
  Week 2: number analyzed (Participants) | 912 | 452
  Week 2 | 1.49 (1.13) | 1.25 (0.93)
  Week 4: number analyzed (Participants) | 903 | 450
  Week 4 | 2.15 (1.27) | 2.13 (1.10)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Change in Hb concentration from baseline to week 1 was analysed using a MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [0.19 to 0.34]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Change in Hb concentration from baseline to week 2 was analysed using a MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [0.19 to 0.38]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 4 Change in Hb concentration from baseline to week 4 was analysed using a MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates; Test type: Superiority; p = 0.1091, Mixed model for repeated measures; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.02 to 0.20]

12. Secondary Outcome: Change in S-ferritin Concentration From Baseline to Weeks 1, 2, 4, and 8
Description: Efficacy
  Change in s-ferritin concentration from baseline to weeks 1, 2, 4, and 8.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: ITT. All randomised subjects.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
ng/mL
  Week 1: number analyzed (Participants) | 940 | 456
  Week 1 | 373.5 (228.9) | 105.7 (79.1)
  Week 2: number analyzed (Participants) | 923 | 449
  Week 2 | 211.8 (152.4) | 169.9 (129.8)
  Week 4: number analyzed (Participants) | 916 | 453
  Week 4 | 98.0 (103.9) | 109.2 (108.7)
  Week 8: number analyzed (Participants) | 912 | 456
  Week 8 | 49.0 (79.7) | 58.7 (104.8)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Change in concentrations of s-ferritin from baseline to week 1 was analysed using a MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 267.7, 95% CI 2-sided [246.3 to 289.0]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Change in concentrations of s-ferritin from baseline to week 2 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 41.7, 95% CI 2-sided [25.6 to 57.8]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 4 Change in concentrations of s-ferritin from baseline to week 4 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p = 0.1150, Mixed model for repeated measures; Mean Difference (Final Values) = -9.0, 95% CI 2-sided [-20.3 to 2.2]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 8 Change in concentrations of s-ferritin from baseline to week 8 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p = 0.0812, Mixed model for repeated measures; Mean Difference (Final Values) = -8.3, 95% CI 2-sided [-17.7 to 1.0]

13. Secondary Outcome: Change in Transferrin Saturation (TSAT) From Baseline to Week 1, 2, 4, and 8
Description: Efficacy
  Changes in transferrin saturation (TSAT) from baseline to week 1, 2, 4, and 8.
  TSAT is the value of serum iron divided by the total iron-binding capacity and the unit is %, which referrers to % of iron-binding sites of transferrin being occupied by iron.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: ITT. All randomised subjects.
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
percentage of saturation
  Week 1: number analyzed (Participants) | 933 | 454
  Week 1 | 16.68 (15.66) | 5.84 (10.52)
  Week 2: number analyzed (Participants) | 913 | 448
  Week 2 | 12.33 (13.46) | 10.58 (12.67)
  Week 4: number analyzed (Participants) | 910 | 451
  Week 4 | 11.63 (12.09) | 11.08 (8.59)
  Week 8: number analyzed (Participants) | 909 | 455
  Week 8 | 9.01 (12.58) | 8.87 (9.03)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Change in TSAT from baseline to week 1 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 11.4, 95% CI 2-sided [10.1 to 12.7]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Change in TSAT from baseline to week 2 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p = 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [1.2 to 3.6]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 4 Change in TSAT from baseline to week 4 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p = 0.0162, Mixed model for repeated measures; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [0.2 to 2.1]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 8 Change in TSAT from baseline to week 8 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, include 95% CIs and corresponding p-value; Test type: Superiority; p = 0.0569, Mixed model for repeated measures; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [0.0 to 1.8]

14. Secondary Outcome: Change in Concentrations of Serum Iron (S-iron) From Baseline to Week 1, 2, 4, and 8
Description: Efficacy
  Changes in the concentrations of serum iron (s-iron) from baseline to week 1, 2, 4, and 8.
Time Frame: Baseline, week 1, 2, 4, and 8
Population: ITT. All randomised subjects.
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
μg/dL
  Week 1: number analyzed (Participants) | 871 | 436
  Week 1 | 63.2 (69.7) | 22.4 (44.4)
  Week 2: number analyzed (Participants) | 855 | 434
  Week 2 | 38.8 (58.1) | 37.0 (51.6)
  Week 4: number analyzed (Participants) | 849 | 435
  Week 4 | 31.2 (49.7) | 35.1 (33.2)
  Week 8: number analyzed (Participants) | 850 | 438
  Week 8 | 24.2 (53.3) | 27.6 (32.7)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Change in s-iron from baseline to week 1 was analysed using a Mixed Model for Repeated Measurement (MMRM) including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, including 95% CIs and corresponding p-value; Test type: Superiority; p < 0.0001, Mixed model for repeated measures; Mean Difference (Final Values) = 43.7, 95% CI 2-sided [38.1 to 49.3]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Change in s-iron from baseline to week 2 was analysed using a Mixed Model for Repeated Measurement (MMRM) including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, including 95% CIs and corresponding p-value; Test type: Superiority; p = 0.0375, Mixed model for repeated measures; Mean Difference (Final Values) = 5.0, 95% CI 2-sided [0.3 to 9.8]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 4 Change in s-iron from baseline to week 4 was analysed using a Mixed Model for Repeated Measurement (MMRM) including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, including 95% CIs and corresponding p-value; Test type: Superiority; p = 0.6027, Mixed model for repeated measures; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-4.0 to 2.3]
Statistical Analysis 4: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 8 Change in s-iron from baseline to week 8 was analysed using a Mixed Model for Repeated Measurement (MMRM) including treatment, week, treatment-by-week interaction, and strata as factors and baseline value and baseline value-by-week interaction as covariates. The estimated treatment differences based on the least square means of the treatment-by-week interaction effects are presented by week, including 95% CIs and corresponding p-value; Test type: Superiority; p = 0.8207, Mixed model for repeated measures; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-2.7 to 3.4]

15. Secondary Outcome: Change in Fatigue Symptoms From Baseline to Week 1, 2, and 8
Description: Efficacy
  Change in fatigue symptoms from baseline to week 1, 2, and 8 was measured by the Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale.
  The Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale consisted of 13 items ranging from 0 (not at all) to 4 (very much), except items #7 and #8 which are reversed scored. The total score range is 0-52.
  A score of less than 30 indicated severe fatigue, and the higher the score, the better outcome/quality of life (QoL). If more than 50% of the items for a subject at a given visit were missing, the total score was not calculated.
  Total score was calculated as shown below:
  Total score= Sum of individual scores x 13 / Number of items answered
Time Frame: Baseline, week 1, 2, and 8
Population: ITT. All randomised subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
score on a scale
  Week 1: number analyzed (Participants) | 940 | 471
  Week 1 | 7.98 (10.41) | 7.38 (9.38)
  Week 2: number analyzed (Participants) | 930 | 462
  Week 2 | 10.74 (11.58) | 11.89 (11.35)
  Week 8: number analyzed (Participants) | 916 | 459
  Week 8 | 14.08 (12.70) | 15.36 (12.87)
Statistical Analysis 1: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 1 Change in fatigue symptoms score from baseline to week 1 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline score and baseline score-by-week interaction as covariates; Test type: Superiority; p = 0.0422, Mixed model for repeated measures; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [0.04 to 2.01]
Statistical Analysis 2: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 2 Change in fatigue symptoms score from baseline to week 2 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline score and baseline score-by-week interaction as covariates; Test type: Superiority; p = 0.4646, Mixed model for repeated measures; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-1.44 to 0.66]
Statistical Analysis 3: Comparison: Iron Isomaltoside/Ferric Derisomaltose vs Iron Sucrose; Week 8 Change in fatigue symptoms score from baseline to week 8 was analysed using MMRM including treatment, week, treatment-by-week interaction, and strata as factors and baseline score and baseline score-by-week interaction as covariates; Test type: Superiority; p = 0.5703, Mixed model for repeated measures; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-1.39 to 0.76]

16. Secondary Outcome: Intervals in Screening for Diabetic Retinopathy (ISDR) Questionnaire, Cost of Public Transport/Taxi And Parking
Description: Pharmacoeconomics
  The Intervals in Screening for Diabetic Retinopathy (ISDR) questionnaire at the baseline visit assessed the resources used by subjects to receive treatment. Resources used on other trial activities were not included. ISDR responses were summarised using descriptive statistics.
  The data for this endpoint show the responses at baseline for both treatment groups.
  The frequency of drug administration between the 2 treatment groups is different, however, (i.e. up to a factor 5 in the iron sucrose treatment group).
Time Frame: Baseline
Population: ITT. All randomised subjects.
Measure: Median (Full Range); unit: US dollars ($)
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
US dollars ($)
  Cost of public transport/taxi: number analyzed (Participants) | 191 | 93
  Cost of public transport/taxi | 5.0 [0 to 52] | 5.0 [0 to 100]
  Cost of parking: number analyzed (Participants) | 789 | 394
  Cost of parking | 0.0 [0 to 30] | 0.0 [0 to 26]

17. Secondary Outcome: Intervals in Screening for Diabetic Retinopathy (ISDR) Questionnaire, Return Journey by Car
Description: as for outcome 16
Time Frame: Baseline
Population: ITT. All randomised subjects.
Measure: Median (Full Range); unit: miles
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 788 | 393
miles | 15.0 [0 to 200] | 15.0 [0 to 120]

18. Secondary Outcome: Intervals in Screening for Diabetic Retinopathy (ISDR) Questionnaire, Time Spent on Visit/Helping on Visit
Description: as for outcome 16
Time Frame: Baseline
Population: ITT. All randomised subjects.
Measure: Median (Full Range); unit: Hours
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
Hours
  Time spent on visit: number analyzed (Participants) | 958 | 479
  Time spent on visit | 2.0 [0.0 to 20.0] | 2.0 [0.2 to 6.8]
  Total time spent helping on visit: number analyzed (Participants) | 195 | 103
  Total time spent helping on visit | 2.0 [0.0 to 8.0] | 2.0 [0.0 to 6.0]

19. Secondary Outcome: Intervals in Screening for Diabetic Retinopathy (ISDR) Questionnaire, Participants/Others Who Took Time Off Work to Attend Visits
Description: as for outcome 16
Time Frame: Baseline
Population: ITT. All randomised subjects.
Measure: Number; unit: participants
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 1009 | 503
participants
  In employment, YES: number analyzed (Participants) | 995 | 496
  In employment, YES | 529 | 258
  Took time off work to attend, YES: number analyzed (Participants) | 529 | 257
  Took time off work to attend, YES | 233 | 113
  Assistance by others to attend visit, YES: number analyzed (Participants) | 997 | 496
  Assistance by others to attend visit, YES | 211 | 111
  Others took time off work to attend, YES: number analyzed (Participants) | 210 | 111
  Others took time off work to attend, YES | 64 | 32

20. Secondary Outcome: Health Care Resource Use Questionnaire
Description: Pharmacoeconomics
  Resources used by the health care staff (per administration), measured by the health care resource use questionnaire. The questionnaire assessed the time used by the health care staff during administration of the investigational product and the administration time (including the observational time). The health care participants included in the evaluation were: investigator, pharmacist, physician, study coordinator, study nurse.
  The data for this endpoint show the responses at baseline for both treatment groups.
  The frequency of drug administration between the treatment groups is different (i.e. up to a factor 5 more frequent in the iron sucrose treatment group).
Time Frame: Baseline
Population: ITT. All randomised subjects.
Measure: Median (Full Range); unit: hours
Groups:
- Iron Isomaltoside/Ferric Derisomaltose: Health care staff involved in the iron isomaltoside/ferric derisomaltose treatment group.
  Assessment of the time used by the health care staff during administration of the investigational product and the administration time (including the observational time).
- Iron Sucrose: Health care staff involved in the iron sucrose treatment group.
  Assessment of the time used by the health care staff during administration of the investigational product and the administration time (including the observational time).
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
Number analyzed (Participants) | 2706 | 1296
hours
  Time spent per site staff median | 1.08 [0.0 to 8.0] | 1.00 [0.0 to 5.5]
  Time spent per subject median: number analyzed (Participants) | 999 | 493
  Time spent per subject median | 3.38 [0.0 to 13.5] | 3.00 [0.0 to 15.8]

ADVERSE EVENTS:
Time Frame: From the time a subjects had signed the informed consent form (CRF) and until they had completed the study, all adverse events (AEs) or serious adverse events (SAEs) were reported in the CRF. The actual study duration was 8 weeks (or shorted if the trial was discontinued). Overall, eligible subjects participated in the trial for approximately 10-15 weeks (including a 14-day screening period and if necessary a run-in period).
Description: AEs were described in a precise, standard medical terminology (i.e. not necessarily the exact words used by the subject). If known, a specific diagnosis was stated. Furthermore, the Investigator assessed an AE regarding seriousness, severity, relatedness, and outcome.
  Of the 1009 subjects in the iron isomaltoside/ferric derisomaltose arm and 503 in the iron sucrose arm, 989 subjects and 494 subjects received treatment, respectively, and were included in the safety population (i.e. at risk).
Arm/Group | Iron Isomaltoside/Ferric Derisomaltose | Iron Sucrose
All-Cause Mortality (participants affected / at risk) | 1/989 | 0/494
Serious Adverse Events (participants affected / at risk) | 21/989 | 13/494
Other Adverse Events (participants affected / at risk) | 31/989 | 16/494
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside/Ferric Derisomaltose (N=989) | Iron Sucrose (N=494)
Abdominal adhesions faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside/Ferric Derisomaltose (N=989) | Iron Sucrose (N=494)
Nausea (Gastrointestinal disorders) | 31 (32) | 16 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution may publish the study results. Before submission for publication or presentation, Institution shall allow Sponsor not less than 90 days to review any manuscript and not less than 30 days to review any poster presentation, abstract, or any other written or oral material which describes or discloses the study results. If sponsor so requests in writing, Institution shall withhold any publication or presentation for an additional 90 days.

DOCUMENTS (2):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT02940886/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT02940886/SAP_001.pdf